CLINICAL TRIAL: NCT00193427
Title: Phase II Trial of Preoperative (Neo-adjuvant) Therapy in Patients With Stages IB, II, IIIA, and Selected IIIB Patients With Non-Small Cell Lung Cancer
Brief Title: Preoperative Therapy in Patients With Stages IB, II, IIIA, and Selected IIIB Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Aventis Pharmaceuticals (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 76
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2012-11-13 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Docetaxel; Gemcitabine; Carboplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Patients with potentially resectable clinical stage IB, II, and selected III NSCLC received gemcitabine 1000 mg/m2 days 1, 8 and docetaxel 30 mg/m2 days 1, 8 every 21 days for 3 cycles. Patients were restaged after treatment and resected 3-6 weeks later. If patients were inoperable, had incomplete resections or N2 disease, docetaxel 20 mg/m2 and carboplatin AUC = 1.5 weekly x 7 and radiation to 63 Gy was administered
  Interventions: Drug: Docetaxel; Drug: Gemcitabine; Drug: Carboplatin; Radiation: Radiation

INTERVENTIONS:
Drug: Docetaxel — 30mg/m2 administered on days 1 and 8, 21-cycle days, 3 cycles
  Other Names: Taxotere
Drug: Gemcitabine — 1000 mg/m2 administered by 30-minute IV infusion on day 1 and 8, 21-cycle days, 3 cycles
  Other Names: Gemzar
Drug: Carboplatin — AUC = 1.5 weekly x 7
  Other Names: Paraplatin
Radiation: Radiation — To 63 Gy

SUMMARY:
This trial is designed to study the role of docetaxel/gemcitabine, an active and relatively non-toxic combination in advanced NSCLC. This study will help to better define optimal preoperative regimens for patients with resectable NSCLC. Since both of these drugs are potent radio-sensitizers, the concurrent use with radiation therapy at these weekly doses may produce not only radio-sensitization, but also considerable antitumor efficacy.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will receive:

Pre-operative

* Docetaxel
* Gemcitabine Post-operative
* Docetaxel
* Carboplatin
* Radiation Therapy

Patients with stage IB and II NSCLC who achieved clear margins will not receive any further therapy. Patients with incomplete resection, resection margins of a T3 tumor that are positive or close, stage IIIA AND IIIB NSCLC or disease judged unresectable after preoperative chemotherapy will receive postoperative treatment

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Histologically confirmed non-small cell lung cancer
* Must be operable candidate
* Clinical stage IB, II, and select III non-small cell lung cancer are eligible
* Measurable or evaluable disease
* Able to perform activities of daily living with minimal assistance
* Must be > 18 years of age
* Adequate bone marrow, liver or kidney
* No previous chemotherapy or radiation therapy for non-small cell lung cancer
* Moderate to severe peripheral neuropathy
* Understand the nature of this study and give written informed consent.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Stage IV disease
* History of prior malignancy within five years
* Women who are pregnant or breast-feeding

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-04; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spigel, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 75
Completed | 26
Not Completed | 49

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 75
Age, Continuous [Median (Full Range); unit: years] | 62 [42 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 47
Region of Enrollment [Number; unit: participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate
Description: A pathological complete response (pCR) was defined as having no residual cancer at the primary site or in regional lymph nodes on pathologic review.
Time Frame: 18 months
Population: All patients who underwent a thoracotomy were assigned a pathologic response category.
Measure: Number; unit: Percentage of participants
Arm/Group | Intervention
Number analyzed (Participants) | 38
Percentage of participants | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival was calculated as the elapsed time between the date of study registration and the date of recurrence or death from any cause.
Time Frame: 19 months
Population: All patients were assessed for progression free survival after a median follow up of 19 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Intervention
Number analyzed (Participants) | 67
Months | 9.9 [5.9 to 13.9]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate is the percentage of patients with complete response or partial response per RECIST v.1 Criteria. Complete response (CR) = Disappearance of all target lesions, disappearance of all nontarget lesions for at least 4 weeks. Partial Response (PR) = At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameters.
Time Frame: 18 months
Population: Patients who were assessable after completion of 9 weeks of treatment were evaluated and assigned a response category.
Measure: Number; unit: percentage of participants
Arm/Group | Intervention
Number analyzed (Participants) | 67
percentage of participants | 30

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was calculated as the elapsed time bewteen date of study registration and the date of death.
Time Frame: 18 months
Population: All patients were assessed for overall survival after a median follow-up of 19 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Intervention
Number analyzed (Participants) | 67
Months | 18 [14.8 to 21.3]

ADVERSE EVENTS:
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 39/75
Other Adverse Events (participants affected / at risk) | 75/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=75)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Cardiac General - Other (Coronary Artery Disease) (Cardiac disorders) | 1
Cardiac ischemia/infarction (Cardiac disorders) | 1
Cardiopulmonary arrest (Cardiac disorders) | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Death not associated with CTCAE term (Death NOS) (General disorders) | 2
Death not associated with CTCAE term (Disease Progression NOS) (General disorders) | 4
Dehydration (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Edema (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Infections and infestations) | 2
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infection - Other (bronchitis) (Infections and infestations) | 1
Infection with normal ANC - Lung (pnemonia) (Infections and infestations) | 1
Infection with unknown ANC - Lung (pnemonia) (Infections and infestations) | 3
Intra-operative injury - Heart (Surgical and medical procedures) | 1
Obstruction, GI - Bowel NOS (Gastrointestinal disorders) | 1
Pulmonary/Upper Respiratory - Other (Acute respiratory failure) (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory - Other (Chronic Obstructive Pulmonary Disease) (Respiratory, thoracic and mediastinal disorders) | 4
Thrombosis/thrombus/embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=75)
Alopecia (Skin and subcutaneous tissue disorders) | 24
Hemoglobin (Blood and lymphatic system disorders) | 50
Anorexia (Gastrointestinal disorders) | 32
Mood alteration - anxiety (Psychiatric disorders) | 6
Pain - joint (Musculoskeletal and connective tissue disorders) | 8
Constipation (Gastrointestinal disorders) | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dehydration (Gastrointestinal disorders) | 8
dysphagia (Gastrointestinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Edema (Blood and lymphatic system disorders) | 11
Esophagitis (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 72
Fever (General disorders) | 5
Hemorrhage, pulmonary/upper respiratory (Blood and lymphatic system disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hypotension (Cardiac disorders) | 5
Infection (Infections and infestations) | 27
Insomnia (General disorders) | 11
Leukocytes (Blood and lymphatic system disorders) | 46
Mucositis (Gastrointestinal disorders) | 10
Pain - muscles (Musculoskeletal and connective tissue disorders) | 5
Nausea (Gastrointestinal disorders) | 36
Neuropathy - sensory (Nervous system disorders) | 6
Neutrophils (Blood and lymphatic system disorders) | 39
Pain (NOS) (General disorders) | 28
Pulmonary Symptoms (Respiratory, thoracic and mediastinal disorders) | 28
Radiation esophagitis (Gastrointestinal disorders) | 14
Skin toxicity (Skin and subcutaneous tissue disorders) | 22
Taste Alteration (Gastrointestinal disorders) | 7
Platelets (Blood and lymphatic system disorders) | 51
Vomiting (Gastrointestinal disorders) | 12
Weight Loss (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.